CLINICAL TRIAL: NCT01017991
Title: Effects of an Infant Formula With Probiotics on Signs and Symptoms of "Colic".
Brief Title: Feeding Intervention for Infants With Crying
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been terminated as a result of low enrollment.
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 09.03.INF
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Crying
Keywords: infants; formula; probiotic; crying
MeSH Terms: conditions — Crying | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infant formula with probiotic (Experimental): Infant formula with probiotic for 0 to 12 months of age
  Interventions: Other: Milk based infant formula with probiotic
- Standard infant formula (Placebo Comparator): Infant formula for 0 to 12 months of age
  Interventions: Other: Milk based infant formula

INTERVENTIONS:
Other: Milk based infant formula with probiotic — formula supplied as a powder to be constituted as commercially available formula ad libitum daily 28 days duration
  Arms: Infant formula with probiotic
Other: Milk based infant formula — supplied as a powder to be constituted as commercially available formula ad libitum daily 28 days
  Arms: Standard infant formula

SUMMARY:
The purpose of the study is to assess if infants who have excessive crying and fussing have less of these symptoms when fed a formula containing a probiotic compared to those fed a standard infant formula.

ELIGIBILITY:
Inclusion Criteria:

* full term infants greater than or equal to 37 wks gestation
* 3 weeks to less than or equal to 4 months of age upon enrollment
* experiencing ongoing crying and fussy episodes of a minimum of 3 hours of crying /day for 3 days in a week for at least one week prior to enrollment
* otherwise healthy as reported by parent/caregiver
* is under the care of a pediatrician or other qualified healthcare professional and has had at least one postnatal visit
* taking no more than one feeding of breast milk per day
* having not initiated weaning foods or beverages other than infant formula or breast milk
* study explained and written information provided with Parent/caregiver demonstrating understanding of the given information
* informed consent signed(parent/legal representative)

Exclusion Criteria:

* Chromosomal or major congenital anomalies
* known cow's milk allergy
* receiving any type of therapeutic formula (including extensively hydrolyzed formula or free amino acid formula)
* receiving an antibiotic or probiotic in the week prior to enrollment
* complicated reflux, defined by reflux combined with inadequate growth and/or respiratory complications
* infant's family, who in the investigator's assessment, cannot be expected to comply with the protocol
* infant currently participating in another conflicting clinical study

Ages: 3 Weeks to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
daily total crying time | 28 days

SECONDARY OUTCOMES:
Formula intake | 4 days
Tolerance evaluated by stool, vomiting, spitting and flatulence frequencies | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Cabana, MD,MPH, Principal Investigator — University of California, San Francisco, USA
Locations (9):
- United States (9):
  - Children's Investigational Research Program, LLC, Bentonville, Arkansas
  - University of California, San Francisco, San Francisco, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Institute for Clinical Research, Orlando, Florida
  - Pedia Research, LLC, Newburgh, Indiana
  - Pedia Research, Owensboro, Kentucky
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Cook Children's Medical Center, Fort Worth, Texas
  - Southwest Children's Research Associates, P.A., San Antonio, Texas